CLINICAL TRIAL: NCT00199693
Title: Hemodynamic and Respiratory Function in Healthy Pregnant Women - A Longitudinal Study
Brief Title: Hemodynamic and Respiratory Function in Healthy Pregnant Women
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Divisiion of Anaethesia and Intensive care medicine, Rikshospitalet, Divisiion of Anaethesia and Intensive care medicine, Rikshospitalet
Other Study IDs: Elangestork2005-1
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2009-06

CONDITIONS: Healthy
Keywords: Hemodynamic and respiratory changes and pregnancy; Healthy pregnant women

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study looks at hemodynamic and respiratory function in healthy pregnant women; it is a longitudinal study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eldrid Langesæter, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Rikshospitalet-Radiumhospitalet HF, Oslo, Norway